CLINICAL TRIAL: NCT00410228
Title: A Single Center, Randomized, Double-Blind, Placebo-and Positive-Controlled, Interleaved, Ascending Single Dose Study to Explore the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AHTT956 in Healthy Subjects
Brief Title: Study to Explore the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AHT956 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAHT956A2101
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: safety, tolerability, pharmacokinetics, pharmacodynamics, AHT956

INTERVENTIONS:
Drug: AHT956

SUMMARY:
This study will evaluate the safety and tolerability of ascending single oral doses of AHT956 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects age 18 to 45 years of age included, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Vital signs must be within the following ranges: oral body temperature between 35.0-37.5 °C; systolic blood pressure, 90-145 mm Hg; diastolic blood pressure, 50-95 mm Hg; pulse rate, 40-90 bpm
* Female subjects must either:have been surgically sterilized or hysterectomized at last 6 months prior to study participation with clinical documentation be postmenopausal (no regular menstrual bleeding for at least 1 year prior to study start)
* Body mass index must be within the range of 18 to 28 kg/m². Subjects must weigh at least 50 kg to participate in this study.

Exclusion Criteria:

* Smokers (any subject who uses tobacco or has cotinine greater than 500 ng/mL)).
* Subjects who received live vaccine 4 weeks prior to dosing, any prescription drug use with 4 weeks prior to dosing, or over-the-counter medication use within 2 weeks prior to dosing.
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing, or longer if required by local regulation.
* Flu-like symptoms or significant within two weeks prior to dosing.
* A past medical history of clinically significant abnormality detected during electrocardiogram (ECG) examination or an evident family history (grandparents, parents and siblings) of a ECG abnormality (i.e. prolonged QT-interval syndrome).
* History of fainting, hypotension when standing up, arrhythmia.
* History of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
* History of clinically significant drug allergy or history of atopic allergy, urticaria, eczematous dermatitis). A known hypersensitivity to the study drugs or drugs similar to the study drugs.
* Any history of surgical or medical condition(s) which could change the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject, including history of gastrointestinal, pancreatic, liver, kidney, bladder, blood, or immune systems.
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted the screening or baseline evaluations.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42
Dates: Start 2006-06

PRIMARY OUTCOMES:
Safety, tolerability of ascending single doses of AHT956 in healthy subjects
MTD (Maximum Tolerated Dose)

SECONDARY OUTCOMES:
Pharmacokinetics of single oral doses of AEB071
Inhibition of T-cell function and lymphocytes proliferation following single rising oral of AHT956
Pharmacokinetic/pharmacodynamic relationship of single rising oral doses of AHT956 at the end of study
Identify gene expression patterns of blood cells

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Bern, Switzerland